CLINICAL TRIAL: NCT02565888
Title: A Drug-drug Interaction Study Between the Novel Anti-HCV Agent Daclatasvir and the Antiretroviral Agents Atazanavir/Ritonavir or Atazanavir/Cobicistat in Healthy Volunteers
Brief Title: A Drug-drug Interaction Study Between Daclatasvir and Atazanavir/Ritonavir or Atazanavir/Cobicistat
Acronym: DATE-4
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: UMCN-AKF 14.12
Record Dates: First submitted 2015-09-30; First posted 2015-10-01 (Estimated); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Hepatitis C; HIV
Keywords: Hepatitis C; HIV; atazanavir; ritonavir; daclatasvir; cobicistat
MeSH Terms: conditions — Hepatitis C | interventions — daclatasvir; Atazanavir Sulfate; Ritonavir; Cobicistat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment A (Active Comparator): Daclatasvir 30 mg QD film-coated tablet + atazanavir 300mg QD hard capsule + ritonavir 100mg QD from film-coated tablet for 10 days.
  Interventions: Drug: Daclatasvir; Drug: Atazanavir; Drug: Ritonavir
- Treatment B (Experimental): Daclatasvir 30 mg QD film-coated tablet + atazanavir 300mg QD hard capsule + cobicistat 150mg QD from film-coated tablet for 10 days.
  Interventions: Drug: Daclatasvir; Drug: Atazanavir; Drug: Cobicistat

INTERVENTIONS:
Drug: Daclatasvir
  Other Names: Daklinza
Drug: Atazanavir
  Other Names: Reyataz
Drug: Ritonavir
  Other Names: Norvir
  Arms: Treatment A
Drug: Cobicistat
  Other Names: Tybost
  Arms: Treatment B

SUMMARY:
This study aims to provide the evidence that 150mg of cobicistat will have the same effect on the pharmacokinetics of daclatasvir 30mg QD as 100mg of ritonavir, when given together with atazanavir 300mg.

DETAILED DESCRIPTION:
Approximately 20-25% of the total number of HIV-infected patients is co-infected with HCV which translates to 6-8 million persons worldwide. Combined treatment of HIV and HCV is complicated by the risk of drug-drug interactions as both the direct acting antiviral agents (DAAs) for HCV as the antiretroviral agents for HIV are substrates of cytochrome P450 (CYP450) or various membrane transporters, and also have the capacity to influence these systems. A careful selection of the appropriate regimens and if needed adjusted doses is key for optimal treatment of both viral infections.

Daclatasvir is a recently approved anti-HCV agent that is a CYP3A4 substrate but does not affect CYP450 itself. It is also a moderate inhibitor of various membrane transporters such as organic anion-transporting polypeptide (OATP1B1), P-glycoprotein (P-gP), and organic cation transporters (OCT2).

Atazanavir/ritonavir is one of the preferred antiretroviral agents in all international guidelines. Ritonavir is used as a boosting agents based on its inhibitory effects on CYP3A. This also inhibits CYP3A-mediated metabolism of daclatasvir and when atazanavir/ritonavir is combined with daclatasvir, it is recommended to reduce the dose of daclatasvir from 60mg QD to 30mg QD.

Cobicistat has recently been approved as an alternative booster of atazanavir at a dose of 150mg QD. It is expected that cobicistat will inhibit CYP3A mediated metabolism of daclatasvir in a similar manner as ritonavir does, but there are no clinical data to support this. As cobicistat lacks some of the adverse events associated with ritonavir use, the use of cobicistat, including as a booster of atazanavir, is likely to increase.

This study aims to provide the evidence that 150mg of cobicistat will have the same effect on the pharmacokinetics of daclatasvir 30mg QD as 100mg of ritonavir, when given together with atazanavir 300mg.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 and not older than 55 years at screening.
2. Subject does not smoke more than 10 cigarettes, 2 cigars, or 2 pipes per day for at least 3 months prior to Day 1.
3. Subject has a Quetelet Index (Body Mass Index) of 18 to 30 kg/m2, extremes included.
4. Subject is able and willing to sign the Informed Consent Form prior to screening evaluations.
5. Subject is in good age-appropriate health condition as established by medical history, physical examination, and electrocardiography, results of biochemistry, hematology and urinalysis testing within 4 weeks prior to day 1. Results of biochemistry, hematology and urinalysis testing should be within the laboratory's reference ranges (see Appendix A). If laboratory results are not within the reference ranges, the subject is included on condition that the Investigator judges that the deviations are not clinically relevant. This should be clearly recorded.
6. Subject has a normal blood pressure and pulse rate, according to the Investigator's judgment.

Exclusion Criteria:

1. Creatinine clearance below 60mL/min.
2. Documented history of sensitivity/idiosyncrasy to medicinal products or excipients.
3. Positive HIV test.
4. Positive hepatitis B or C test.
5. Pregnant female (as confirmed by an hCG test performed less than 4 weeks before day 1) or breast-feeding female. Female subjects of childbearing potential without adequate contraception, e.g. hysterectomy, bilateral tubal ligation, (non-hormonal) intrauterine device, total abstinence, double barrier methods, or two years post-menopausal. They must agree to take precautions in order to prevent a pregnancy throughout the entire conduct of the study.
6. Therapy with any drug (for two weeks preceding Day 1), except for acetaminophen (max 2 gram/day).
7. Relevant history or presence of pulmonary disorders (especially COPD), cardiovascular disorders, neurological disorders (especially seizures and migraine), psychiatric disorders, gastro-intestinal disorders, renal and hepatic disorders (clinically relevant increased ALAT/ASAT or hyperbilirubinemia) hormonal disorders (especially diabetes mellitus), coagulation disorders.
8. Relevant history or current condition that might interfere with drug absorption, distribution, metabolism or excretion.
9. History of or current abuse of drugs, alcohol or solvents.
10. Inability to understand the nature and extent of the study and the procedures required.
11. Participation in a drug study within 60 days prior to Day 1.
12. Donation of blood within 60 days prior to Day 1.
13. Febrile illness within 3 days before Day 1.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
AUC | up to 24 hours after administration

SECONDARY OUTCOMES:
Adverse events | 4 weeks
  adverse events will be collected up to 4 weeks in total (entire study)

CONTACTS AND LOCATIONS:
Overall Officials: David Burger, PharmD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- CRCN, Radboud University Medical Center, Nijmegen, Netherlands

REFERENCES:
- [Result] Smolders EJ, Colbers EP, de Kanter CT, Velthoven-Graafland K, Drenth JP, Burger DM. Daclatasvir 30 mg/day is the correct dose for patients taking atazanavir/cobicistat. J Antimicrob Chemother. 2017 Feb;72(2):486-489. doi: 10.1093/jac/dkw429. Epub 2016 Oct 20. PMID 27798211
- [Derived] Overbeek JK, van Erp NP, Burger DM, den Broeder AA, Koolen SLW, Huitema ADR, Ter Heine R. Population Pharmacokinetics of Cobicistat and its Effect on the Pharmacokinetics of the Anticancer Drug Olaparib. Clin Pharmacokinet. 2025 Mar;64(3):425-435. doi: 10.1007/s40262-025-01480-w. Epub 2025 Feb 5. PMID 39909979